CLINICAL TRIAL: NCT01235429
Title: Specific Aim 3: Partners in Care Randomized Controlled Trial
Brief Title: Partners in Care Diabetes Self-management Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Joseph K Kaholokula, Department of Native Hawaiian Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PILI ARRA Supplement
Record Dates: First submitted 2010-11-03; First posted 2010-11-05 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Behavioral intervention; diabetes self-management; Native Hawaiians; health disparities
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational (Experimental): Participants will receive 12 diabetes self-management educational lessons in a small group setting located within the participating communities and delivered by trained community health workers.
  Interventions: Behavioral: Partners in Care
- Delayed education (Active Comparator): The delayed education group will receive the same intervention after the intervention group has completed the educational lessons and all participants have completed the follow-up assessments.
  Interventions: Behavioral: Partners in Care

INTERVENTIONS:
Behavioral: Partners in Care — Participants will be offered 12 group diabetes self-management educational lessons delivered by trained community health workers.
  Arms: Educational
Behavioral: Partners in Care — Diabetes self-management education
  Arms: Delayed education

SUMMARY:
Type 2 diabetes is common among Native Hawaiians and Pacific Peoples. Diabetes related complications decrease quality of life and can result in early morbidity. The purpose of the Partners in Care diabetes self-management educational intervention is to teach participants how to manage their diabetes to avoid or delay diabetes-related complications and how to better work with their health care team.

DETAILED DESCRIPTION:
This is a feasibility study using a randomized controlled trial (RCT) design in which 100 Native Hawaiians (NHs) and other Pacific Islanders (PPs) will be randomized to either a 3-month diabetes self-management group (DSMG; N=50) or a delayed intervention control group (CG; N=50). Participants in the DSMG will receive culturally-tailored, group diabetes self-management education delivered in a community setting by trained community peer educators. To meet this objective, we have partnered with four community-based organizations: 1) Hawai'i Maoli Association of Hawaiian Civic Clubs, 2) Ke Ola Mamo Native Hawaiian Health Care System, 3) Kokua Kalihi Valley Comprehensive Family Services, and 4) Kula No Nā Po'e Hawai'i. These four organizations provide services to a large number of Pacific People to include, but not limited to, Native Hawaiians, Samoans, Filipinos, and Chuukese. They already have intervention research experience as members of the PILI 'Ohana CBPR Project. The 3-month face-to-face intervention will be community-based and community-led by trained community peer educators from these four partnering community organizations. Individuals with a hemoglobin A1c (HbA1c; average blood sugar levels) >=8% will be recruited for the study because they represent the most at-risk for diabetes-related complications.

Over a 1-year accrual period, the community partners will recruit and enroll 100 eligible NHs and PPs (25 participants per a participating community), as well as deliver and evaluate the intervention in their respective community settings. The primary outcomes of our study are hemoglobin A1c and self-reported diabetes specific quality of life. Secondary outcomes are cholesterol levels (including HDL, LDL, total cholesterol, and triglycerides), blood pressure, body mass index, and psychosocial adaptation.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported Native Hawaiian, Filipino, or other Pacific Islander ethnic background,
2. Adults age >=18 years,
3. English-speaking,
4. Physician-diagnosed type 2 diabetes, and
5. Baseline hemoglobin A1c >=8%

Exclusion Criteria:

1. Survival less than 6 months,
2. Planning to move off island or out of state during the study period,
3. Pregnancy,
4. Any co-morbid condition (physical and mental disabilities) that would prevent the individual from participating in the intervention protocol (i.e., major psychiatric illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c | 3 months
  Hemoglobin A1c will be assessed at baseline and post intervention in the intervention and delayed intervention participants.

SECONDARY OUTCOMES:
Quality of life | 3 months
  Quality of life using the Problem Areas in Diabetes survey will be assessed at baseline and post intervention in the intervention and delayed intervention participants.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Kaholokula, PhD, Principal Investigator — University of Hawaii
Locations (1):
- University of Hawaii, Honolulu, Hawaii, United States